CLINICAL TRIAL: NCT02614248
Title: The Use of Coconut Oil for the Prevention and Treatment of Diaper Dermatitis in the NICU Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genesis Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 817035
Record Dates: First submitted 2015-11-16; First posted 2015-11-25 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Dermatitis, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coconut Oil (Experimental): Participants in this group will receive a generous layer of organic, unrefined coconut oil applied to the diaper area (buttocks and creases between thighs and hips) at each diaper change. This will continue until the patient is discharged or reaches the primary safety endpoint (skin that is eroded and/or blistered in the diaper area with bleeding).
  Interventions: Other: Organic, Unrefined Coconut Oil
- Standard of Care (Active Comparator): Participants in this group will receive the standard of care for preventing and treating diaper dermatitis at Genesis. This includes no treatment until a diaper dermatitis appears. If diaper dermatitis appears, participants will receive a generous layer of Medline Remedy Phytoplex Z-Guard Skin Protectant applied to the diaper area (buttocks and creases between thighs and hips) at each diaper change. This will continue until the patient is discharged or reaches the primary safety endpoint (skin that is eroded and/or blistered in the diaper area with bleeding).
  Interventions: Other: Medline Remedy Phytoplex Z-Guard Skin Protectant

INTERVENTIONS:
Other: Organic, Unrefined Coconut Oil
  Arms: Coconut Oil
Other: Medline Remedy Phytoplex Z-Guard Skin Protectant
  Arms: Standard of Care

SUMMARY:
The purpose of the study is to examine the safety and effectiveness of the use of coconut oil for the prevention and treatment of diaper dermatitis among NICU babies at Genesis Medical Center, Davenport.

ELIGIBILITY:
Inclusion Criteria:

1. Babies admitted to the Genesis NICU
2. Anticipated stay in the NICU is ≥ 48 hours
3. Babies wearing diapers 24 hours a day
4. Parent willing to sign informed consent for the study
5. Parent willing to use the test products in the diaper area during the trial
6. Parent willing to not change the type or brand of diaper and wipes during the study
7. Parent willing to refrain from changing any other products whose use may have an effect of their baby's skin condition during the trial

Exclusion Criteria:

1. Babies with a gestational age <30 weeks
2. Babies with major congenital malformations
3. Active dermatological conditions other than diaper dermatitis that may affect trial results
4. Known sensitivity to ingredients in trial products
5. Babies whose parents have a hazelnut or coconut allergy
6. Other severe acute medical conditions that may increase the risk associated with trial participation

Ages: 5 Hours to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Genesis Medical Center, East Campus, Davenport, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Coconut Oil: Participants in this group will receive a generous layer of organic, unrefined coconut oil applied to the diaper area (buttocks and creases between thighs and hips) at each diaper change. This will continue until the patient is discharged or reaches the primary safety endpoint (skin that is eroded and/or blistered in the diaper area with bleeding).
  Organic, Unrefined Coconut Oil
- Standard of Care: Participants in this group will receive the standard of care for preventing and treating diaper dermatitis at Genesis. This includes no treatment until a diaper dermatitis appears. If diaper dermatitis appears, participants will receive a generous layer of Medline Remedy Phytoplex Z-Guard Skin Protectant applied to the diaper area (buttocks and creases between thighs and hips) at each diaper change. This will continue until the patient is discharged or reaches the primary safety endpoint (skin that is eroded and/or blistered in the diaper area with bleeding).
  Medline Remedy Phytoplex Z-Guard Skin Protectant
Period: Overall Study
Arm/Group | Coconut Oil | Standard of Care
Started | 75 | 74
Completed | 72 | 70
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coconut Oil | Standard of Care | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 74 | 149
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Days] | 3.0 [1 to 71] | 3.0 [1 to 77] | 3.0 [1 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 43 | 46 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 74 | 149

OUTCOME MEASURES:

1. Primary Outcome: The Number of Days Free From Diaper Dermatitis
Description: The number of days free from diaper dermatitis.
Time Frame: Once, at hospital discharge, an average of 2 weeks
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Coconut Oil | Standard of Care
Number analyzed (Participants) | 75 | 74
Days | 4.065 (0) | 4.274 (0)

2. Primary Outcome: The Number of Patients Experiencing Adverse Events
Description: The number of patients experiencing adverse events.
Time Frame: Once, at hospital discharge, an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Coconut Oil | Standard of Care
Number analyzed (Participants) | 75 | 74
Participants | 29 | 22

3. Secondary Outcome: The Percent of Parents Stating Satisfaction With the Diaper Dermatitis Treatment Used
Description: The percent of parents stating satisfaction with the diaper dermatitis treatment used Measured by a parent satisfaction survey
Time Frame: Once, at study completion for hospital discharge, an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Coconut Oil | Standard of Care
Number analyzed (Participants) | 66 | 65
Participants | 60 | 55

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Coconut Oil | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 29/75 | 23/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coconut Oil (N=75) | Standard of Care (N=74)
Respiratory syncitial virus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lingual frenum (General disorders) | 1 (1) | 1 (1)
Neonatal hyperbilirubinemia (Hepatobiliary disorders) | 6 (6) | 8 (8)
Localized eruption of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash on back- not diaper rash
Bleeding skin (Skin and subcutaneous tissue disorders) | 20 (20) | 13 (13) — Diaper area bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT02614248/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02614248/SAP_001.pdf